CLINICAL TRIAL: NCT05672758
Title: The Effect of Long-lasting Adaptation to Intensive Speed-power and Endurance Training on Plasma Free Amino Acids Concentration at Rest, During Graded Exercise and Post-exercise Recovery
Brief Title: Effect of Long-lasting Adaptation to Endurance and Speed-power Training on Plasma Free Amino Acids Concentration
Acronym: AAdaptation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of Medical Sciences (Other); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Krzysztof Kusy, Associated Professor, Poznan University of Physical Education
Other Study IDs: OPUS 14 2017/27/B/NZ7/02828
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Healthy Athletes Aged 18-35 Years
Keywords: free plasma amino acids; competitive athletes; sprint training; endurance training; mass spectrometry
MeSH Terms: interventions — High-Intensity Interval Training; Endurance Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sprint-Trained Athletes: Highly trained track sprinters at the national or international level aged 18-35 years with sport experience 5-10 years; structured periodized training
  Interventions: Behavioral: Sprint training
- Endurance-Trained Athletes: Highly trained long-distance runners and triathletes at the national or international level aged 18-35 years with sport experience 5-10 years; structured periodized training
  Interventions: Behavioral: Endurance training
- Amateur/Recreational Athletes (Controls): Individuals participating in amateur non-professional sport aged 18-35 years with activity experience 5-10 years; unstructured non-periodized training
  Interventions: Behavioral: Recreational Training

INTERVENTIONS:
Behavioral: Sprint training — One-year cycle including specific sprint-oriented athletic training
  Groups: Sprint-Trained Athletes
Behavioral: Endurance training — One-year cycle including specific endurance-oriented athletic training
  Groups: Endurance-Trained Athletes
Behavioral: Recreational Training — One year of nonspecific recreational training
  Groups: Amateur/Recreational Athletes (Controls)

SUMMARY:
The goal of this observational study was to detect the long-term effect of two different training modalities - speed-power and endurance training - on changes in plasma free amino acid (PFAA) concentration at rest, during graded exercise and post-exercise recovery period. It was assumed that these training modalities cause different amino acids concentration in human blood depending on long-term sport specialization and predominant exercise type (the contribution of high-intensity exercise related to anaerobic metabolism). The hypotheses were:

1. highly-trained speed-power have higher concentrations of PFAA than endurance athletes;
2. PFAA concentration varies with the change in training loads in a one-year training cycle. Higher PFAA concentrations is expected in training phases with larger contribution of high-intensity exercise;
3. PFAA concentration per 1 kg muscle mass differ between speed-power and endurance athletes.

Forty-eght highly-trained athletes aged 18-32 years with longer competitive sport experience - sprinters vs triathletes/distance runners - and 10 recreationally trained controls were examined. Laboratory tests were conducted in consecutive training subphases.

(i) Body composition and muscle mass was assessed using densitometry. (ii) Participants underwent a graded exercise treadmill test until exhaustion. (iii) Blood samples were drawn at rest, during exercise (every 3 min, at each speed change), and after exercise (immediately and 5, 10, 15, 20 and 30 min post exercise).

(iv)The analysis of PFAA profiles was based on the Liquid Chromatography Electrospray Ionization tandem Mass Spectrometry (LC-ESI-MS/MS) technique and the aTRAQ reagent. This allowed to quantify 42 PFAAs.

The results improve the understanding of metabolic adaptation to long-term exercise programmes. Possible practical application encompasses the domains of exercise medicine, sport and public health.

The novelty of the project: (1) comparing the effect of two different training models on PFAA concentration, (2) tracking the changes in PFAAs across a one-year training cycle, (3) repeated multiple sampling in one exercise session including resting conditions, (4) introducing skeletal muscle mass as a factor potentially affecting PFAA profiles, (5) a large number (42) of proteinogenic- and non-proteinogenic PFAAs, (6) homogenous highly-trained athletic groups, and (7) a proven state-of-the-art method to determine PFAAs.

DETAILED DESCRIPTION:
I. Study goal

Long-term effect of two different training modalities - speed-power and endurance training - on changes in plasma free amino acid (PFAA) concentration at rest, during graded exercise until exhaustion and recovery period was compared. The model cohorts were highly-trained athletes. The assumption was that structured long-lasting speed-power and endurance training cause adaptations resulting in different PFAA concentration and that the changes depend on long-term sport specialization (predominant exercise type) and training phase of the one-year cycle (contribution of high-intensity exercise based on anaerobic metabolism characterized by rapid adenosine-5'-triphosphate degradation). A larger contribution of high-intensity exercise is used by speed-power athletes and in phases of specific preparation/competition. There is a lack of research on long-term effects of physical training on changes in PFAAs. This picture is supllemented by monitoring changes in a set of 42 proteinogenic and non-proteinogenic PFAAs. Short- and long-lasting effects of training on levels and time course of PFAA concentration during exercise and recovery will be shown. The main goals were:

1. To compare the effect of the two entirely different training modalities (speed-power and endurance) on PFAA concentration.
2. To observe the effect of training load character on changes in resting, exercise and post-exercise PFAA concentration in consecutive training phases of a one-year training cycle.
3. To determine the link between PFAA concentration and exercise modality, taking into account skeletal muscle mass.

II. Background

Only 3-6% of the total energy utilized during prolonged endurance exercise is derived from oxidation of AAs. However, the proportion of energy from AA catabolism considerably increases during exercise. Although protein turnover does not contribute substantially to the energy expenditure, it may fill other important functions during exercise. AAs may delay muscle glycogen depletion.

The free AA pool amounts only 2% of the total AA amount and is stored within the plasma and intra- and extracellular spaces. This small pool accounts for a continuous exchange of AAs. Blood plasma serves as a temporary reservoir of AAs, the size of which changes in response to exercise. Differences in regular training, exercise, and daily activities result in differences in PFAA levels.

Exercise duration affects PFAA levels, however, the direction of the changes may be different for specific AAs and exercise type, intensity, and duration. In contrast, muscle AAs concentration remains relatively stable. AA metabolism during prolonged exercise has been described. Reports based on a short training periods (few weeks) in power-type athletes suggest that sprint and endurance training sessions have a distinct effect on serum AAs. However, there is a lack of studies on the differences in long-term adaptation changes in PFAAs between endurance- and sprint-trained individuals, taking into account multiple blood sampling (rest, exercise, recovery) and muscle mass.

III. Methods

Over 70 athletes aged 18-32 years - speed-power (sprinters), endurance (triathletes, distance runners), and recreationally trained - were recruited. Eventually, the data of 58 of them were considered for analysis. Athletes were examined four times during one-year training cycle: (1) general preparation phase, (2) specific preparation phase, (3) competition phase, and (4) transition phase.

The main statistical tool was one-way and two-way ANOVA with repeated measures. The required sample size was computed based on given alpha (significance) level, statistical power, and effect size. The significance level α < 0.05 and statistical power 0.8 were assumed. Based on earlier studies that compared sprint- and endurance-trained athletes in terms of other metabolic phenomena related to training and exercise, minimum partial eta square (η2) of 0.2 was adopted, i.e. a large effect size for differences between examined groups and consecutive examination across was expected. Other assumptions were nonsphericity correction = 0.75, number of measurements = 4, and correlation between repeated measurements = 0.5. The minimum total sample size of 22 athletes was obtained.

Body composition was assessed using dual X-ray absorptiometry (Lunar Prodigy, GE Healthcare, USA). Skeletal muscle mass was estimated using regression equations.

Graded exercise tests on a treadmill (h/p/cosmos, Germany) were conducted before 12 a.m., two hours after a standard meal. The initial speed was 8 km/h and increased every 3 min by 2 km/h until exhaustion. Respiratory parameters and heart rate were measured (ergospirometer MetaLyzer 3B, Cortex, Germany; Polar Elektro RS 400, Finland). Maximum oxygen consumption was measured.

Blood sampling. Peripheral venous catheter was placed into dorsal metacarpal vein. Blood samples were drawn at rest, during exercise (every 3 min, at each speed change), and immediately, 5, 10, 15, 20, and 30 min after exercise completion. The volume of venous blood obtained during one examination was 25 ml, i.e. 2.5 ml for each sample, up to 10 samples. Each sample was collected into plasma-separation tube containing EDTA for further plasma analysis. Samples were centrifuged at 13,000 revolution/min for 3 min at 4°C. Obtained plasma was then pipetted into 0.5 ml vials and immediately frozen in liquid nitrogen. Samples were stored in -80°C until analysis.

Forty two PFAAs were assayed: O-Phospho-L-serine, O-Phosphoethanolamine, Taurine, L-Asparagine, L-Serine, Hydroxy-L-proline, Glycine, L-Glutamine, Ethanolamine, L-Aspartic acid, L-Citrulline, Sarcosine, β-Alanine, L-Alanine, L-Threonine, L-Glutamic acid, L-Histidine, 1-Methyl-L-histidine, 3-Methyl-L-histidine, L-Homocitrulline, Argininosuccinic acid, γ-Amino-n-butyric acid, D, L-β-Aminoisobutyric acid, L-α-Amino-n-butyric acid, L- α- Aminoadipic acid, L-Anserine, L-Carnosine, L-Proline, L-Arginine, δ-Hydroxylysine, L-Ornithine, Cystathionine, L-Cystine, L-Lysine, L-Valine, L-Methionine, L-Tyrosine, L-Homocystine, L-Isoleucine, L-Leucine, L-Phenylanine, L-Tryptophan. The analysis of PFAAs was based on the LC-ESI-MS/MS technique and the aTRAQ (Sciex) reagent, characterized by high sensitivity and specificity, short analytical run time, low sample volume required to perform the analysis, and high amount of analytes being quantified in one run.

Protocol for determination of PFAAs. Plasma samples of 40 µl were transferred to Eppendorf tubes. In order to precipitate proteins present in plasma, 10 µl of 10% sulfosalicylic acid was added and the content was mixed and centrifuged (10,000 g for 2 minutes). After that, the supernatant was transferred to a new tube and mixed with 40 µl of borate buffer. An aliquot of 10 µl of the obtained solution was subsequently labeled with the aTRAQ reagent Δ8 solution (5 µl), mixed, centrifuged, and incubated at room temperature for 30 minutes. The labeling reaction was then stopped by addition of 5 µl of 1.2% hydroxylamine, mixed, and incubated at room temperature for 15 minutes. After that, 32 µl of the internal standard solution was added and the content was mixed. In the next step, the sample was evaporated in a vacuum concentrator for 15 minutes to reduce the volume of the sample to about 20 µl. The residue was then diluted with 20 µl of water, mixed, and transferred to an autosampler vial with an insert. This procedure was modified in order to measure the concentrations of PFAAs that could not be detected using the original method. For this purpose, plasma samples of higher volume were used for the sample preparation procedure. Instead of 40 μl, plasma samples of 80 μl were transferred to Eppendorf tubes and mixed with 20 μl of 10% sulfosalicylic acid. After that, 20 μl of the supernatant was transferred to a new tube and mixed with 30 μl of borate buffer. The subsequent steps of the procedure remained unchanged. The internal standard solution contained the same AAs labeled with the aTRAQ reagent Δ0. Thus, each determined PFAA had its corresponding internal standard. Norleucine and norvaline, two non-proteinogenic AAs, were used to evaluate the labeling efficiency and recovery. Their corresponding internal standards were also present in the internal standard solution.

The analyses were performed using the liquid chromatography instrument 1260 Infinity (Agilent Technologies) coupled to the 4000 QTRAP (quadrupole ion trap) mass spectrometer (Sciex). This mass spectrometer is equipped with an electrospray ionization source and three quadrupoles and allows to conduct the quantitative PFAA analysis planned within the presented project. The chromatographic separation was performed with the Sciex C18 (5 μm, 4.6 mm x 150 mm) chromatography column. The flow rate of mobile phases was maintained at 800 μl/min. The method uses the following mobile phases: water (phase A) and methanol (phase B), both with addition of 0,1 % formic acid and 0.01 % heptafluorobutyric acid. The time of analysis was 18 minutes and during that time the chromatographic separation was carried out with the following gradient elution: from 0 till 6 min - from 2% to 40% of phase B, then maintained at 40% of phase B for 4 minutes, increased to 90% of phase B till 11 min and held at that ratio phases for 1 minute, then decreased to 2% of phase B and finally maintained at 2% of phase B from 13 to 18 min. The injection volume was set at 2 μl and the separation temperature at 50 °C. The ion source settings were the following: curtain gas 20 psig; ion spray voltage 4500 V; ion source temperature 600 °C; ion source gas 1 = 60 psig, ion source gas 2 = 50 psig. The mass spectrometer operated in positive ionization mode and the following parameters were applied: entrance potential = 10 V; declustering potential = 30 V; collision cell exit potential = 5 V; collision energy = 30 eV (50 eV in case of 7 compounds); collision gas: nitrogen. The PFAAs were measured in scheduled multiple reaction monitoring (sMRM) mode. This mode ensures high specificity and sensitivity in quantitative analyses. A system suitability test (analysis of a standard mixture of AAs) was conducted before each batch of samples in order to warm up and check the inter-day performance of the whole system. Data acquisition and processing were performed using the Analyst 1.5 software (Sciex). The described LC-ESI-MS/MS method for determination of AAs is well established in the Department of Inorganic and Analytical Chemistry, Poznan University of Medical Sciences, the co-investigator of the project.

Total blood count was performed using the device Mythic 18 (Orphée, Swiss). Capillary blood samples from fingertip (20 μl per sample) were drawn simultaneously with venous blood pre-, during and postexercise. Blood lactate concentration was measured using C-line analyzer (EKF-Diagnostic, Germany).

ELIGIBILITY:
Inclusion Criteria for professional athletes:

* highly trained sprint- and endurance-trained athletes
* national or international performance level
* current participation in training programs organized by professional sports clubs or national team (licence) for at least 5 years
* current medical eligibility for competitive sport

Inclusion Criteria for amateur/recreational athletes:

* regular recreational activity for at least 5 years (preferred endurance disciplines)
* participation in amateur competition
* good health status
* non-smoking

Exclusion Criteria for professional athletes:

* untrained individuals
* athletes that do not meet the above criteria for participation in professional sport
* injured athletes or those who are not able or willing to participate for other reasons

Exclusion Criteria for amateur/recreational athletes:

* inactive/sedentary individuals
* medical contraindications to high-intensity exercise and testing
* injured individuals or those who are not able or willing to participate for other reasons
* current smokers or heavy past smokers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Highly trained competitive athletes aged 18-35 years with longer competitive sport experience, specialized in sports of different character - speed-power (sprinters) vs endurance (triathletes, distance runners). Amateur/recreational athletes participating in training on a regular basis.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
absolute Plasma Free Amino Acids Concentration (42 amino acids) | 4 times in a 1-year training cycle: at rest, during graded exercise (every 3 min), and during recovery (5, 10, 15, 20, and 30 min)
  µmol/L
relative Plasma Free Amino Acids Concentration (42 amino acids) | 4 times in a 1-year training cycle: at rest, during graded exercise (every 3 min), and during recovery (5, 10, 15, 20, and 30 min)
  µmol/L/kg muscle mass

SECONDARY OUTCOMES:
absolute Skeletal Muscle Mass (aSMM) | 4 times in a 1-year training cycle
  kg
relative Skeletal Muscle Mass (rSMM) | 4 times in a 1-year training cycle
  percent of total body mass
absolute Lean Body Mass (aLBM) | 4 times in a 1-year training cycle
  kg
relative Lean Body Mass (rLBM) | 4 times in a 1-year training cycle
  percent of total body mass
absolute Fat Mass (aFM) | 4 times in a 1-year training cycle
  kg
relative Fat Mass (rFM) | 4 times in a 1-year training cycle
  percent of total body mass
absolute Maximum Oxygen Uptake (aVO2max) | 4 times in a 1-year training cycle
  L/min
relative Maximum Oxygen Uptake 1 (r1VO2max) | 4 times in a 1-year training cycle
  L/min/kg total body mass
relative Maximum Oxygen Uptake 2 (r2VO2max) | 4 times in a 1-year training cycle
  L/min/kg skeletal muscle mass

OTHER OUTCOMES:
White Blood Cells | 4 times in a 1-year training cycle
  10^9/L
Red Blood Cells | 4 times in a 1-year training cycle
  10^12/L
Hematocrit | 4 times in a 1-year training cycle
  percent
Mean Corpuscular Volume (MCV) | 4 times in a 1-year training cycle
  fL
Mean Corpuscular Hemoglobin (MCH) | 4 times in a 1-year training cycle
  pg
Mean Corpuscular Hemoglobin Concentration (MCHC) | 4 times in a 1-year training cycle
  g/dL
Red Blood Cell Volume Distribution Width (RDW-CV) | 4 times in a 1-year training cycle
  percent
Blood Lactate Concentration | 4 times in a 1-year training cycler: at rest, during graded exercise (every 3 min), and during recovery (5, 10, 15, 20, and 30 min)
  mmol/L
Blood Ammonia | 4 times in a 1-year training cycle: at rest, during graded exercise (every 3 min), and during recovery (5, 10, 15, 20, and 30 min)
  µmol/L
Creatine Kinase at rest | 4 times in a 1-year training cycle
  U/L
Maximum Heart Rate (HRmax) | 4 times in a 1-year training cycle
  beats per min
Appendicular Lean Soft Tissue (ALST) | 4 times in a 1-year training cycle
  kg
Relative Skeletal Muscle Mass Index (RSMI) | 4 times in a 1-year training cycle
  kg/m^2
Weight | 4 times in a 1-year training cycle
  kg
Height | 4 times in a 1-year training cycle
  kg
Body Mass Index (BMI) | 4 times in a 1-year training cycle
  kg/m^2
Age | baseline
  years
Sports History (Experience) | baseline
  years
Speed at VO2max (vVO2max) | baseline
  km/h
Maximum Minute Ventilation (VEmax) | 4 times in a 1-year training cycle
  L/min
Maximum Tidal Volume (VT) | 4 times in a 1-year training cycle
  L
Maximum Breathing Frequency (BF) | 4 times in a 1-year training cycle
  /min

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Kusy, PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Wielkoolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 1 year after publication of the data
Access Criteria: Scientists specialized in amino acids and training research on request (kusy@awf.poznan.pl). Principal investigator will review the requests

REFERENCES:
- [Background] Ahlborg G, Felig P, Hagenfeldt L, Hendler R, Wahren J. Substrate turnover during prolonged exercise in man. Splanchnic and leg metabolism of glucose, free fatty acids, and amino acids. J Clin Invest. 1974 Apr;53(4):1080-90. doi: 10.1172/JCI107645. PMID 4815076
- [Background] Ahlborg G, Felig P. Lactate and glucose exchange across the forearm, legs, and splanchnic bed during and after prolonged leg exercise. J Clin Invest. 1982 Jan;69(1):45-54. doi: 10.1172/jci110440. PMID 7054242
- [Background] Areces F, Gonzalez-Millan C, Salinero JJ, Abian-Vicen J, Lara B, Gallo-Salazar C, Ruiz-Vicente D, Del Coso J. Changes in Serum Free Amino Acids and Muscle Fatigue Experienced during a Half-Ironman Triathlon. PLoS One. 2015 Sep 15;10(9):e0138376. doi: 10.1371/journal.pone.0138376. eCollection 2015. PMID 26372162
- [Background] Ballard FJ, Tomas FM. 3-Methylhistidine as a measure of skeletal muscle protein breakdown in human subjects: the case for its continued use. Clin Sci (Lond). 1983 Sep;65(3):209-15. doi: 10.1042/cs0650209. No abstract available. PMID 6872455
- [Background] Blomstrand E, Celsing F, Newsholme EA. Changes in plasma concentrations of aromatic and branched-chain amino acids during sustained exercise in man and their possible role in fatigue. Acta Physiol Scand. 1988 May;133(1):115-21. doi: 10.1111/j.1748-1716.1988.tb08388.x. PMID 3227900
- [Background] Borgenvik M, Nordin M, Mikael Mattsson C, Enqvist JK, Blomstrand E, Ekblom B. Alterations in amino acid concentrations in the plasma and muscle in human subjects during 24 h of simulated adventure racing. Eur J Appl Physiol. 2012 Oct;112(10):3679-88. doi: 10.1007/s00421-012-2350-8. Epub 2012 Feb 18. PMID 22350359
- [Background] Castell LM, Newsholme EA. Glutamine and the effects of exhaustive exercise upon the immune response. Can J Physiol Pharmacol. 1998 May;76(5):524-32. doi: 10.1139/cjpp-76-5-524. PMID 9839078
- [Background] Cuisinier C, Ward RJ, Francaux M, Sturbois X, de Witte P. Changes in plasma and urinary taurine and amino acids in runners immediately and 24h after a marathon. Amino Acids. 2001;20(1):13-23. doi: 10.1007/s007260170062. PMID 11310927
- [Background] Decombaz J, Reinhardt P, Anantharaman K, von Glutz G, Poortmans JR. Biochemical changes in a 100 km run: free amino acids, urea, and creatinine. Eur J Appl Physiol Occup Physiol. 1979 Apr 12;41(1):61-72. doi: 10.1007/BF00424469. PMID 446472
- [Background] Derezinski P, Klupczynska A, Sawicki W, Palka JA, Kokot ZJ. Amino Acid Profiles of Serum and Urine in Search for Prostate Cancer Biomarkers: a Pilot Study. Int J Med Sci. 2017 Jan 1;14(1):1-12. doi: 10.7150/ijms.15783. eCollection 2017. PMID 28138303
- [Background] Einspahr KJ, Tharp G. Influence of endurance training on plasma amino acid concentrations in humans at rest and after intense exercise. Int J Sports Med. 1989 Aug;10(4):233-6. doi: 10.1055/s-2007-1024908. PMID 2606590
- [Background] Felig P, Wahren J. Amino acid metabolism in exercising man. J Clin Invest. 1971 Dec;50(12):2703-14. doi: 10.1172/JCI106771. PMID 5129318
- [Background] Gibala MJ. Regulation of skeletal muscle amino acid metabolism during exercise. Int J Sport Nutr Exerc Metab. 2001 Mar;11(1):87-108. doi: 10.1123/ijsnem.11.1.87. PMID 11255139
- [Background] Graham TE, Turcotte LP, Kiens B, Richter EA. Training and muscle ammonia and amino acid metabolism in humans during prolonged exercise. J Appl Physiol (1985). 1995 Feb;78(2):725-35. doi: 10.1152/jappl.1995.78.2.725. PMID 7759446
- [Background] Hajduk J, Klupczynska A, Derezinski P, Matysiak J, Kokot P, Nowak DM, Gajecka M, Nowak-Markwitz E, Kokot ZJ. A Combined Metabolomic and Proteomic Analysis of Gestational Diabetes Mellitus. Int J Mol Sci. 2015 Dec 16;16(12):30034-45. doi: 10.3390/ijms161226133. PMID 26694367
- [Background] Haralambie G, Berg A. Serum urea and amino nitrogen changes with exercise duration. Eur J Appl Physiol Occup Physiol. 1976 Dec 6;36(1):39-48. doi: 10.1007/BF00421632. PMID 1001315
- [Background] Hargreaves MH, Snow R. Amino acids and endurance exercise. Int J Sport Nutr Exerc Metab. 2001 Mar;11(1):133-45. doi: 10.1123/ijsnem.11.1.133. PMID 11255141
- [Background] Hassmen P, Blomstrand E, Ekblom B, Newsholme EA. Branched-chain amino acid supplementation during 30-km competitive run: mood and cognitive performance. Nutrition. 1994 Sep-Oct;10(5):405-10. PMID 7819652
- [Background] Henriksson J. Effect of exercise on amino acid concentrations in skeletal muscle and plasma. J Exp Biol. 1991 Oct;160:149-65. doi: 10.1242/jeb.160.1.149. PMID 1960512
- [Background] Huq F, Thompson M, Ruell P. Changes in serum amino acid concentrations during prolonged endurance running. Jpn J Physiol. 1993;43(6):797-807. doi: 10.2170/jjphysiol.43.797. PMID 8007448
- [Background] Ishikura K, Miyakawa S, Yatabe Y, Takekoshi K and Ohmori H. Effect of taurine supplementation on blood glucose concentration during prolonged exercise. Tairyoku Kagaku (Japanese Journal of Physical Fitness and Sport Medicien). 2008; 57, 475-484. [in Japanese]
- [Background] Kim J, Wang Z, Heymsfield SB, Baumgartner RN, Gallagher D. Total-body skeletal muscle mass: estimation by a new dual-energy X-ray absorptiometry method. Am J Clin Nutr. 2002 Aug;76(2):378-83. doi: 10.1093/ajcn/76.2.378. PMID 12145010
- [Background] Kim J, Shen W, Gallagher D, Jones A Jr, Wang Z, Wang J, Heshka S, Heymsfield SB. Total-body skeletal muscle mass: estimation by dual-energy X-ray absorptiometry in children and adolescents. Am J Clin Nutr. 2006 Nov;84(5):1014-20. doi: 10.1093/ajcn/84.5.1014. PMID 17093152
- [Background] Klupczynska A, Derezinski P, Dyszkiewicz W, Pawlak K, Kasprzyk M, Kokot ZJ. Evaluation of serum amino acid profiles' utility in non-small cell lung cancer detection in Polish population. Lung Cancer. 2016 Oct;100:71-76. doi: 10.1016/j.lungcan.2016.04.008. Epub 2016 May 7. PMID 27597283
- [Background] Lemon PW, Mullin JP. Effect of initial muscle glycogen levels on protein catabolism during exercise. J Appl Physiol Respir Environ Exerc Physiol. 1980 Apr;48(4):624-9. doi: 10.1152/jappl.1980.48.4.624. PMID 7380688
- [Background] Matysiak J, Derezinski P, Klupczynska A, Matysiak J, Kaczmarek E, Kokot ZJ. Effects of a honeybee sting on the serum free amino acid profile in humans. PLoS One. 2014 Jul 29;9(7):e103533. doi: 10.1371/journal.pone.0103533. eCollection 2014. PMID 25072247
- [Background] Newsholme EA, Leech TR. Functional biochemistry in health and disease. Wiley-Blackwell, Chichester 2010.
- [Background] Pitkanen H, Mero A, Oja SS, Komi PV, Pontinen PJ, Saransaari P, Takala T. Serum amino acid responses to three different exercise sessions in male power athletes. J Sports Med Phys Fitness. 2002 Dec;42(4):472-80. PMID 12391443
- [Background] Pitkanen H, Mero A, Oja SS, Komi PV, Rusko H, Nummela A, Saransaari P, Takala T. Effects of training on the exercise-induced changes in serum amino acids and hormones. J Strength Cond Res. 2002 Aug;16(3):390-8. PMID 12173953
- [Background] Rennie MJ, Edwards RH, Krywawych S, Davies CT, Halliday D, Waterlow JC, Millward DJ. Effect of exercise on protein turnover in man. Clin Sci (Lond). 1981 Nov;61(5):627-39. doi: 10.1042/cs0610627. PMID 7285508
- [Background] Tarnopolsky M. Protein requirements for endurance athletes. Nutrition. 2004 Jul-Aug;20(7-8):662-8. doi: 10.1016/j.nut.2004.04.008. PMID 15212749
- [Background] Wagenmakers AJ. Muscle amino acid metabolism at rest and during exercise: role in human physiology and metabolism. Exerc Sport Sci Rev. 1998;26:287-314. PMID 9696993
- [Background] Ward RJ, Francaux M, Cuisinier C, Sturbois X, De Witte P. Changes in plasma taurine levels after different endurance events. Amino Acids. 1999;16(1):71-7. doi: 10.1007/BF01318886. PMID 10078335
- [Background] Wolfe RR, Wolfe MH, Nadel ER, Shaw JH. Isotopic determination of amino acid-urea interactions in exercise in humans. J Appl Physiol Respir Environ Exerc Physiol. 1984 Jan;56(1):221-9. doi: 10.1152/jappl.1984.56.1.221. PMID 6420382
- [Background] Xiao Q, Moore SC, Keadle SK, Xiang YB, Zheng W, Peters TM, Leitzmann MF, Ji BT, Sampson JN, Shu XO, Matthews CE. Objectively measured physical activity and plasma metabolomics in the Shanghai Physical Activity Study. Int J Epidemiol. 2016 Oct;45(5):1433-1444. doi: 10.1093/ije/dyw033. Epub 2016 Apr 12. PMID 27073263
- [Background] Zielinski J, Kusy K. Training-induced adaptation in purine metabolism in high-level sprinters vs. triathletes. J Appl Physiol (1985). 2012 Feb;112(4):542-51. doi: 10.1152/japplphysiol.01292.2011. Epub 2011 Dec 8. PMID 22162524